CLINICAL TRIAL: NCT04928391
Title: Optic Nerve Sheath Diameter (ONSD): A New Modality to Assess Postoperative Agitation After a Single Bolus of Dexmedetomidine Versus Normal Saline in Children With Cleft Palate Repair
Brief Title: A Single Bolus of Dexmedetomidine Versus Normal Saline in Postoperative Agitation
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300616
Record Dates: First submitted 2021-06-10; First posted 2021-06-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cleft Palate
MeSH Terms: conditions — Cleft Palate | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Experimental): Dexmedetomidine IV at the end of surgery
  Interventions: Drug: Dexmedetomidine
- Group C (Placebo Comparator): Same volume of saline placebo IV at the end of surgery
  Interventions: Other: 0.9% saline

INTERVENTIONS:
Drug: Dexmedetomidine — A single dose of 0.5 µ/kg IV dexmedetomidine at the end of surgery
  Other Names: Precedex
  Arms: Group D
Other: 0.9% saline — Same volume of saline placebo IV at the end of surgery
  Other Names: Normal saline
  Arms: Group C

SUMMARY:
The hypothesis of this study is to investigate and compare the efficacy between the administrations of single intravenous (IV) dose of dexmedetomidine versus normal saline in preventing immediate postoperative agitation in children undergoing cleft palate repair.

DETAILED DESCRIPTION:
A written informed consent will be taken from the guardian of children.Patients will be assigned randomly to three groups (30 subjects each) to be anesthetized. The study drug will be delivered in opaque bags labeled "study drug" and 90 patients will be allocated in three groups (of 30 patients each) to receive the study drug at the end of surgery; a single dose of 0.5 µ/kg IV dexmedetomidine (Group D) or same volume of saline placebo (Group C).

ELIGIBILITY:
Inclusion Criteria:

* Children (age 1-7 years) of American Society of Anaesthesiologists physical status (ASA) I-II
* Elective cleft palate repair ± cleft lip surgery under general anesthesia.

Exclusion Criteria:

* Ventriculo-peritoneal shunt
* Suspected meningitis
* Congenital hydrocephalus
* Clinical signs of suspected increased intracranial pressure
* On treatment for seizures or metabolic diseases
* Children with developmental delay
* Hypersensitivity to dexmedetomidine or nalbuphine

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-06-20 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
the Pediatric Anesthesia Emergence Delirium (PAED) score | 1 hour postoperative
  Emergence delirium (ED) will be measured by the Pediatric Anesthesia Emergence Delirium (PAED) scale. The scores for each of the five listed behaviours (The child makes eye contact with the caregiver/parent, the child's actions are Purposeful, the child is aware of his/her surroundings, the child is restless and the child is inconsolable) are added to achieve a total score (maximum score of 20). A score of ≥ 12 yields 100% sensitivity and 94.5% specificity for the diagnosis of ED

SECONDARY OUTCOMES:
FLACC (Face, Legs, Activity, Cry, and Consolability) pain score. | 1 hour postoperative
  The FLACC is a behavioural pain assessment scale for use for non-verbal or pre-verbal patients unable to self-report their level of pain. Rate your child in each of the five measurement categories, add together, and document total pain score (0 - 10), score 0= relaxed and no pain, 1-3= mild pain/discomfort, 4-6= moderate pain, 7-10= severe discomfort/pain.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Soliman, Study Director — Assiut University
Locations (2):
- Egypt (2):
  - Omar Soliman, Asyut, Assuit
  - Assiut university hospital, Asyut

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Milic M, Goranovic T, Knezevic P. Complications of sevoflurane-fentanyl versus midazolam-fentanyl anesthesia in pediatric cleft lip and palate surgery: a randomized comparison study. Int J Oral Maxillofac Surg. 2010 Jan;39(1):5-9. doi: 10.1016/j.ijom.2009.09.007. Epub 2009 Oct 24. PMID 19854614